CLINICAL TRIAL: NCT03600090
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of hLAG-3 Fusion Protein, EOC202 (Eftilagimod Alpha) Combined With Paclitaxel in Chinese Patients With Metastatic Breast Cancer
Brief Title: Phase I Study of EOC202 Plus Paclitaxel in Chinese Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taizhou EOC Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EOC202A1101
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-02

CONDITIONS: Solid Tumor, Adult
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm EOC202 + Paclitaxol (Experimental): Biological: EOC202 This study is an open label, non-randomized, fixed dose-escalation phase I study, performed in ambulatory setting with patients receiving as a first line chemotherapy for metastatic breast carcinoma the standard 6 cycles of paclitaxel (80 mg/m² at D1, D8 and D15 of every 4-week cycle).
  Two EOC202 dose levels (6 mg and 30 mg) will be evaluated in two cohorts of 18 patients. At any given dose level the patients will be administered one dose every two weeks for a total of 48 weeks (12 s.c. injections in total), separated by 13-day intervals free of EOC202 administration.
  The repeated single doses will be administered on D2 and D16 of the 4-week cycles, on the day which follows chemotherapy.
  Interventions: Biological: EOC202; Drug: Paclitaxel

INTERVENTIONS:
Biological: EOC202 — EOC202 will be SC injection.
Drug: Paclitaxel — Paclitaxol will be IV injection

SUMMARY:
Open label, single arm, dose-escalation phase I study in ambulatory patients receiving first line chemotherapy for metastatic breast cancer. The treatment comprises of the standard 6 cycles of weekly paclitaxel (80 mg/m² IV at D1, D8 and D15 of a 28 day cycle) and two EOC202 doses (6 and 30 mg SC at D2 and D16 of a 28 day cycle) for 6 cycles. After completion of the combined therapy, the patients can continue to receive up to 6 cycles of EOC202 maintenance monotherapy (once every cycle on day 1 of each cycle).

DETAILED DESCRIPTION:
This study is an open label, single arm, dose-escalation phase I study, performed in ambulatory setting with patients receiving first line chemotherapy for metastatic breast carcinoma. The standard 6 cycles of paclitaxel (80 mg/m² at D1, D8 and D15 of every 4-week cycle) will be given to subjects. Twenty mg i.v. dexamethasone will be given in the first cycle before each paclitaxel infusion. Corticosteroids will not be administered after the first chemotherapy cycle if the first 3 i.v. infusions of paclitaxel have been well tolerated.

Two EOC202 dose levels, 6 mg and 30 mg will be given to subjects during the cycle and be evaluated in successive cohorts of patients. For each dose level, 3 patients will be administered one subcutaneous dose every 2 weeks for a total of 24 weeks (12 injections in total), separated by 13-day administration-free intervals.

The 30 mg dose will be dosed to 3 new patients if the 6 mg dose has been deemed safe and well tolerated.

Cohort A - 3 patients at the 6 mg dose - will receive EOC202 administration in seriatim separated by four-week intervals for DLT observation. If safety/tolerability are acceptable at the end of the DLT observation periods, the study will proceed to the next dose.

Cohort B - 3 patients at the 30 mg dose - will receive EOC202 administration in seriatim separated by four-week intervals for DLT observation. If safety/tolerability are acceptable at the end of the 4-week observation periods, the study will proceed to the next phase.

Cohort C will comprise of additional 6 patients as the PK dose expansion group based on the recommended dose for expansion (RDE). The study procedure is the same with the corresponding dose group.

All patients will participate in a pharmacokinetic (PK) and pharmacodynamic (PD) study which involves additional blood samples.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be able to understand and willing to sign the informed consent form, and to complete the trial procedure and follow-up examinations;
2. Female patients with histologically or cytologically confirmed metastatic breast cancer;
3. Patients with HER-2 negative, including hormone receptor (HR) positive/HER-2 negative and triple negative breast cancer (TNBC);
4. Age 18-70 years (including the critical value);
5. Patients who are judged by investigators as suitable to receive paclitaxel first-line chemotherapy;
6. All female patients with childbearing potential must have a negative highly sensitive pregnancy test within 7 days prior to the first dose of investigational product, and as judged by investigators, will not breastfeed and be willing to use effective contraceptive measures during the trial and at least 6 months after the last dose;
7. ECOG performance status 0 or 1;
8. Expected survival longer than 6 months;
9. The previous adjuvant chemotherapy, targeted therapy, antitumor traditional Chinese medicine or Chinese drug preparation, radiotherapy or surgery prior to the first dose must have been completed for at least 4 weeks, endocrine therapy must have been completed for at least 2 weeks; and all the relevant toxicities (except for alopecia and other adverse events that are judged by investigators as tolerable) have been recovered to grade 1 or normal level.
10. At least one measurable lesion as defined by RECISTV 1.1 evaluation criteria for solid tumors;
11. Good organ function level; 1) Hematology: total white blood cell count ≥ 3x109/L; absolute neutrophil count (ANC) ≥ LLN(lower limit of normal), platelet count ≥ LLN, hemoglobin ≥ 9g/dL; 2) Liver: serum total bilirubin ≤ 1.5 upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤ 3xULN(for patients with Gilbert syndrome, total bilirubin≤ 3xULN is allowed; for patients with hepatic metastasis , total bilirubin ≤ 3xULN, AST and ALT≤ 5xULN are allowed); 3) Renal: serum creatinine ≤ 1.5 x ULN.

Exclusion Criteria:

1. Previous chemotherapy for metastatic breast cancer;
2. Patients with recurrence of breast cancer within 6 months after the last dose of previous adjuvant chemotherapy;
3. Inability to discontinue CYP isoenzyme inhibitor or inducer prohibited in the protocol 2 weeks before the first dose and during the trial;
4. Patients with symptomatic central nervous system metastases;
5. Abnormality on HBV serum tests (5 items) and HBV-DNA (+), anti-HCV antibody (+), HCV-RNA (+), anti-HIV antibody (+), or other serious infection requiring systemic therapy within 4 weeks prior to the first dose of investigational product;
6. Clinically significant ECG abnormality, including but not limited to serious arrhythmia, prolonged QTc (QTcF≥470ms, QTcF=QT/RR0.33), or existence of various factors that may increase the risk of prolonged QTc (hypokalemia, congenital long QT syndrome, or current use of any drug that is known to prolong QTc));
7. Serious or uncontrolled (NYHA III-IV) heart disease within 6 months prior to the first dose of investigational product, including myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, symptomatic congestive heart failure; or presence of cerebrovascular accident, transient ischemic attack, symptomatic pulmonary embolism;
8. History of autoimmune disease, immunodeficiency disease or organ transplantation (including allogeneic bone marrow transplantation), or previous hematopoietic stem cell rescue following chemotherapy, or having active autoimmune disease, immunodeficiency disease, or the disease requiring systemic steroid hormone (>10mg daily prednisone or equivalent dose to 10mg prednisone) or immunomodulatory drug for continuous treatment;
9. Other malignant tumors other than breast cancer in the past three years (except successfully treated squamous cell carcinoma of the skin, superficial bladder cancer, and in situ carcinoma of the cervix);
10. Previous allergy to macromolecular protein preparation or protein, or Quincke's edema (also known as angioneurotic edema), or known allergy to any component of the investigational product, including cremophor EL;
11. History of clear mental disorder, or history of psychotropic drug abuse, drug addiction or alcohol abuse;
12. Vaccination with live attenuated vaccine within 4 weeks prior to the first dose of investigational product, or expected vaccination with live attenuated vaccine during the trial or within 3 months after the end of combined therapy;
13. Previous use of systemic immunomodulator prior to the first dose of investigational product, and discontinuation of the systemic immunomodulator ≤ 5 half-lives of the drug at the first dose;
14. Receiving therapy in any other clinical trial within 4 weeks prior to the first dose of investigational product;
15. Patients who are judged by investigators as unsuitable to participate in the clinical trial as participation in the trial may increase the risk or there may be other severe, acute or chronic disease that may interfere with the interpretation of the trial results;
16. Patients who are not suitable to participate in the trial for other reasons, as judged by investigators.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2021-12-25 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
DLT | From the initiation of protocol treatment to the occurrence of any of the following events: disease progression or disease recurrence or death from any cause, assessed up to 12 months
  DLT and its incidence at each dose level

SECONDARY OUTCOMES:
PFS | up to 24 months
  Progression-free Survival
Cmax | The time points for blood collection are prior to administration of EOC202 on Day 2 of Cycle 1and Day 2 of Cycle 4 and 1h, 2h, 4h, 8h, 24h, 48h, 72h, 144h, 192h
  Maximum Plasma Concentration
Tmax | The time points for blood collection are prior to administration of EOC202 on Day 2 of Cycle 1and Day 2 of Cycle 4 and 1h, 2h, 4h, 8h, 24h, 48h, 72h, 144h, 192h
  Time at which maximum plasma concentration was observed
AUC 0-inf | The time points for blood collection are prior to administration of EOC202 on Day 2 of Cycle 1and Day 2 of Cycle 4 and 1h, 2h, 4h, 8h, 24h, 48h, 72h, 144h, 192h
  Area under the plasma concentration-time curve from time zero to infinity
T1/2 | The time points for blood collection are prior to administration of EOC202 on Day 2 of Cycle 1and Day 2 of Cycle 4 and 1h, 2h, 4h, 8h, 24h, 48h, 72h, 144h, 192h
  Elimination Half-life

OTHER OUTCOMES:
Pharmacodynamic Biomarker | Up to 12 months
  Absolute primary target cells (monocyte (CD14+/CD45+) and dendritic cells (CD45+/HLA-DR+/BDCA-1+ or CD45+/HLA-DR+/BDCA-2+), secondary target cells (CD8+ T cell (CD3+/CD8+) and NK cells (CD3-/CD16+/CD56+)) count and percentage; CCL-4(MIP-1β), IFN-γ, TNF-α, CA125 and CA153 levels in peripheral blood
Immunogenicity Biomarkers | Combined therapy period: prior to administration of paclitaxel on Day 1 of Cycle 1, 2 , 3, 5 (28 day cycle); maintenance monotherapy period: prior to administration of EOC202 on Day1 of Cycle 1, 4 (28 day cycle)
  ADA, ANA and RF

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No